CLINICAL TRIAL: NCT01518517
Title: Phase 2/3 Study Evaluating Efficacy and Safety of Erythrocytes Encapsulating L-asparaginase (GRASPA)Versus Reference L-asparaginase Treatment in Combination With Standard Polychemotherapy in Patient With First Recurrence of Philadelphia Negative Acute Lymphoblastic Leukemia
Brief Title: GRASPA (Erythrocytes Encapsulating L-asparaginase) in Patients With Relapse of Acute Lymphoblastic Leukemia
Acronym: GRASPIVOTALL
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: ERYtech Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GRASPALL2009-06
Record Dates: First submitted 2012-01-10; First posted 2012-01-26 (Estimated); Results first posted 2022-02-02 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-02

CONDITIONS: Acute Lymphoblastic Leukemia, in Relapse
Keywords: acute lymphoblastic leukemia; relapse; asparaginase
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence | interventions — Asparaginase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GRASPA (Experimental): Each patient randomized in GRASPA® group is to receive at least 2 and up to 10 administration of GRASPA® 150 IU/kg, in combination with standard chemotherapy (COOPRALL).
  GRASPA® administration takes place as below:
  * for induction phase: at Day 4 and D18 (F1-F2 induction ) or at D6 if Vanda induction applies (according disease severity)
  * for consolidation phase: at Day 6 of R2 / R1 blocks, each time block of chemotherapy is given (up to 8 cycles)
  Interventions: Drug: GRASPA
- reference L-asparaginase (Active Comparator): For patient randomized in control group, reference L-asparaginase 10,000 IU/m² will be administered every 3 days intravenously, in combination with standard chemotherapy (COOPRALL).
  •for induction phase:at Day 4 , D7, D10, D13 (F1 block ) then at Day 18, D21, D24, D27 (of F2 Blocks).
  NB: administrations take place at D6, D9, D12 and D15 in case of F1-F2 Induction is replaced by VANDA (according disease severity)
  •for consolidation phase: at D6, D9, D12 ofR2/R1 blocks, each time block of chemotherapy is given (up to 8 cycles).
  Interventions: Drug: L-asparaginase

INTERVENTIONS:
Drug: GRASPA — one injection of GRASPA 150 IU/kg at each cycle of chemotherapy
  Other Names: ERY001
  Arms: GRASPA
Drug: L-asparaginase — 3 to 4 Injections of Native E.coli asparaginase 10000IU/m² (every 3 days) at each cycle of chemotherapy
  Other Names: KIDROLASE
  Arms: reference L-asparaginase

SUMMARY:
Asparaginase is a cornerstone in the treatment of ALL, but its utility is limited by toxicities including hypersensitivity. Clinical allergy is associated with inactivation of asparaginase by antibodies (A-Abs), which can also neutralize asparaginase without any clinical signs of hypersensitivity (silent inactivation). GRASPA improves pharmacokinetics, tolerability and maintain circulating asparaginase activity due to the protective barrier of the erythrocyte membrane.

This study is run to confirm the benefit/risk profile of GRASPA at 150 IU/kg in combination with the COOPRALL regimen in adults and children patients with relapsed ALL, with or without known hypersensitivity to L-asparaginase.

DETAILED DESCRIPTION:
This open, randomized international Phase 2/3 study will enrol patients with relapsed ALL. The co-primary endpoints were the duration of asparagine depletion < 2µmol/L and the incidence of asparaginase hypersensitivity during induction. Key secondary endpoints are complete remission (CR), minimal residual disease (MRD), event free survival (EFS) and overall survival (OS).The study was powered to detect 3-fold difference in the incidence of allergic reactions between treatments. patients will be randomized to GRASPA or to Reference L-asparaginase. Patients with history of hypersensitivity to previous L-asparaginase treatment will be treated with GRASPA (exploratory arm)

ELIGIBILITY:
Inclusion Criteria:

* Patient from 1 to 55 years old (Children and adolescents from 1 to 17 years/ Adults from 18 to 55 years)
* Patients with 1st ALL relapse, which could be either isolated bone marrow relapse, or combined (medullary and extra-medullary) relapse, or extra-medullary isolated relapse; or lymphoblastic lymphoma (excepted Burkitt lymphoma) OR Failure to ALL first line treatment (no complete remission obtained)
* Patient previously treated with free E.Coli L-asparaginase form or pegylated one
* Performance Status ≤ 2 (WHO score)
* Patient informed and consent provided (the 2 parents need to consent when children are below 18)

Exclusion Criteria:

* ALL t(9;22) and/or BCR-ABL positive (Philadelphia chromosome positive)
* Patient with 2nd relapse and over
* Women of childbearing potential without effective contraception as well as pregnant or breast feeding women
* Patient unable to receive treatments used in global chemotherapy protocols, due to general or visceral conditions such as:Severe cardiac impairment (NYHA grade 3 or 4 cardiomyopathy)/Serum creatinine 2 x ULN unless related to ALL /ALT or AST 5 x ULN unless related to ALL /Pancreatitis history /Other malignancy that ALL / Severe Infection, HIV positive, active hepatitis related to B or C virus infection / Trisomy 21 / Other serious conditions according to investigator's opinion
* Known grade 4 allergic reaction to E.Coli L-asparaginase (according NCI-CTCAE, Version 3.0)
* History of grade 3 transfusional incident
* Presence of specific anti-erythrocyte antibodies preventing from getting a compatible erythrocyte concentrate for the patient
* Patient under concomitant treatment likely to cause hemolysis
* Patient undergoing yellow fever vaccination
* Patient under phenytoin treatment
* Patient included in previous clinical study less than 6 weeks ago

Ages: 1 Year to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 85 (Actual)
Dates: Start 2009-12 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yves Bertand, MD, Principal Investigator
Locations (28):
- Belgium (2):
  - Hopital Des Enfants Reine Fabiola, Brussels
  - Chr de La Citadelle, Liège
- France (26):
  - Chu D'Angers, Angers
  - Hopital Saint Jacques, Besançon
  - Hopital Pellegrin Enfants, Bordeaux
  - Chu Estaing, Clermont-Ferrand
  - Hopital Henri Mondor, Créteil
  - Chu Grenoble, Grenoble
  - Chru Lille - Hop Jeanne de Flandres, Lille
  - Institut Hematologie Oncologie Pediatrique, Lyon
  - Institut Paoli Calmettes, Marseille
  - Hopital Mere Enfant, Nantes
  - Hotel Dieu, Nantes
  - Hopital de L'Archet 2, Nice
  - Hopital Armand Trousseau, Paris
  - Hopital Robert Debre, Paris
  - Hopital Saint Louis, Paris
  - Hopital Haut-Leveque, Pessac
  - Hopital Lyon Sud, Pierre-Bénite
  - Chru Hopital Sud, Rennes
  - Centre Henri Becquerel, Rouen
  - Chu Hopital Nord, Saint-Etienne
  - Institut Cancerologie de La Loire, Saint-Priest-en-Jarez
  - Hopital de Hautepierre, Strasbourg
  - Chu de Toulouse Enfants, Toulouse
  - Hotel Dieu, Valenciennes
  - Hopital Brabois Enfants, Vandœuvre-lès-Nancy
  - Hopital de Brabois, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- GRASPA (Non Allergic Population); GRASPA (Allergic Population): Each patient randomized in GRASPA® group is to receive at least 2 and up to 10 administration of GRASPA® 150 IU/kg, in combination with standard chemotherapy (COOPRALL).
  GRASPA® administration takes place as below:
  * for induction phase: at Day 4 and D18 (F1-F2 induction ) or at D6 if Vanda induction applies (according disease severity)
  * for consolidation phase: at Day 6 of R2 / R1 blocks, each time block of chemotherapy is given (up to 8 cycles)
  GRASPA: one injection of GRASPA 150 IU/kg at each cycle of chemotherapy
- Reference L-asparaginase (Non Allergic Population): For patient randomized in control group, reference L-asparaginase 10,000 IU/m² will be administered every 3 days intravenously, in combination with standard chemotherapy (COOPRALL).
  •for induction phase:at Day 4 , D7, D10, D13 (F1 block ) then at Day 18, D21, D24, D27 (of F2 Blocks).
  NB: administrations take place at D6, D9, D12 and D15 in case of F1-F2 Induction is replaced by VANDA (according disease severity)
  •for consolidation phase: at D6, D9, D12 ofR2/R1 blocks, each time block of chemotherapy is given (up to 8 cycles).
  L-asparaginase: 3 to 4 Injections of Native E.coli asparaginase 10000IU/m² (every 3 days) at each cycle of chemotherapy
Period: Overall Study
Arm/Group | GRASPA (Non Allergic Population) | Reference L-asparaginase (Non Allergic Population) | GRASPA (Allergic Population)
Started | 29 | 30 | 26
Completed | 1 | 3 | 0
Not Completed | 28 | 27 | 26

BASELINE CHARACTERISTICS:
Groups:
- Reference L-asparaginase (Non Allergic Population: For patient randomized in control group, reference L-asparaginase 10,000 IU/m² will be administered every 3 days intravenously, in combination with standard chemotherapy (COOPRALL).
  •for induction phase:at Day 4 , D7, D10, D13 (F1 block ) then at Day 18, D21, D24, D27 (of F2 Blocks).
  NB: administrations take place at D6, D9, D12 and D15 in case of F1-F2 Induction is replaced by VANDA (according disease severity)
  •for consolidation phase: at D6, D9, D12 ofR2/R1 blocks, each time block of chemotherapy is given (up to 8 cycles).
  L-asparaginase: 3 to 4 Injections of Native E.coli asparaginase 10000IU/m² (every 3 days) at each cycle of chemotherapy
- Total: Total of all reporting groups
Arm/Group | GRASPA (Non Allergic Population) | Reference L-asparaginase (Non Allergic Population | GRASPA (Allergic Population) | Total
Number analyzed (Participants) | 29 | 30 | 26 | 85
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 23 | 23 | 15 | 61
  Between 18 and 65 years | 6 | 7 | 11 | 24
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 8 | 29
  Male | 18 | 20 | 18 | 56

OUTCOME MEASURES:

1. Primary Outcome: Duration of Asparaginase Activity >100 U/L During Induction
Description: Co-primary efficacy endpoint: duration in days of asparaginase activity >100 U/L in whole blood during the induction treatment phase: last available date/time of activity >100 UI/L before activity drops below 100 U/L - date/time of first activity >100 UI/L. Asparaginase activity is compared for GRASPA versus native ASNase to demonstrate the non-inferiority of GRASPA.
Time Frame: Induction treatment period (i.e. 28 days)
Population: Only non allergic population evaluated for efficacy (i.e. 2 randomized arms). Only patient receiving treatment are considered.
Measure: Mean (95% Confidence Interval); unit: days
Groups:
- GRASPA Non Allergic: Each patient randomized in GRASPA® group is to receive at least 2 and up to 10 administration of GRASPA® 150 IU/kg, in combination with standard chemotherapy (COOPRALL).
  GRASPA® administration takes place as below:
  * for induction phase: at Day 4 and D18 (F1-F2 induction ) or at D6 if Vanda induction applies (according disease severity)
  * for consolidation phase: at Day 6 of R2 / R1 blocks, each time block of chemotherapy is given (up to 8 cycles)
  GRASPA: one injection of GRASPA 150 IU/kg at each cycle of chemotherapy
- Reference L-asparaginase: For patient randomized in control group, reference L-asparaginase 10,000 IU/m² will be administered every 3 days intravenously, in combination with standard chemotherapy (COOPRALL).
  •for induction phase:at Day 4 , D7, D10, D13 (F1 block ) then at Day 18, D21, D24, D27 (of F2 Blocks).
  NB: administrations take place at D6, D9, D12 and D15 in case of F1-F2 Induction is replaced by VANDA (according disease severity)
  •for consolidation phase: at D6, D9, D12 ofR2/R1 blocks, each time block of chemotherapy is given (up to 8 cycles).
  L-asparaginase: 3 to 4 Injections of Native E.coli asparaginase 10000IU/m² (every 3 days) at each cycle of chemotherapy
Arm/Group | GRASPA Non Allergic | Reference L-asparaginase
Number analyzed (Participants) | 26 | 28
days | 18.9 [16.7 to 21.0] | 8.5 [6.0 to 11.1]

2. Primary Outcome: Allergic Reaction During Induction Phase
Description: Co-primary safety endpoint: allergic reaction regardless of grade during induction phase. Only those reactions that were reported in relation to the treatment to which the patient was randomised were counted.
Time Frame: Induction treatment period (i.e. 28 days)
Population: Only patient receiving treatment are considered.
Measure: Number; unit: reactions
Arm/Group | GRASPA (Non Allergic Population) | Reference L-asparaginase (Non Allergic Population) | GRASPA (Allergic Population)
Number analyzed (Participants) | 26 | 28 | 26
reactions | 0 | 13 | 3

3. Secondary Outcome: Complete Remission (CR)
Description: CR is defined as, no physical evidence of leukemia, normal CBC, cytologic remission: normally regenerating bone marrow, with <5% leukemic blasts and the absence of detectable CNS or extramedullary disease, evaluated with physical examination and CSF findings, at the end of induction
Time Frame: Induction treatment period (i.e. 28 days)
Measure: Count of Participants; unit: Participants
Arm/Group | GRASPA (Non Allergic Population) | Reference L-asparaginase (Non Allergic Population) | GRASPA (Allergic Population)
Number analyzed (Participants) | 25 | 28 | 25
Participants | 19 | 13 | 15

4. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from randomisation or date of inclusion (allergic arm) until death due to any cause. Patients who did not die were censored at 36 months of follow-up or the date of the patient's last visit, whichever was earlier.
Time Frame: Overall trial period to 36 months
Population: Entries given below are number of patients dying in each group
Measure: Count of Participants; unit: Participants
Arm/Group | GRASPA (Non Allergic Population) | Reference L-asparaginase (Non Allergic Population) | GRASPA (Allergic Population)
Number analyzed (Participants) | 26 | 28 | 26
Participants | 9 | 12 | 14

5. Secondary Outcome: Event Free Survival
Description: EFS is defined as the time from randomisation until the first documented sign of disease relapse or death due to any cause. In line with CHMP guidance (CHMP, 2016), patients who did not achieve CR at the end of the induction period were considered to have had an event at time 0. For the patients enrolled in the GRASPA allergic arm, EFS is defined from the date of inclusion in the study.
  Patients who achieved CR at the end of induction and who did not have a documented relapse or death due to any cause were censored at 36 months of follow-up or the date of the patient's last visit, whichever was earlier.
Time Frame: Overall trial period to 36 months
Population: Entries below are the numbers of patients with events in each treatment group
Measure: Count of Participants; unit: Participants
Arm/Group | GRASPA (Non Allergic Population) | Reference L-asparaginase (Non Allergic Population) | GRASPA (Allergic Population)
Number analyzed (Participants) | 26 | 28 | 26
Participants | 15 | 17 | 19

ADVERSE EVENTS:
Time Frame: AEs were collected from the first trial related activity after the subject signs the informed consent and until 4 months after last dose of study drug depending on the number of doses of asparaginase patients received (depending on study drug exposure period, with a maximum of 1.5 months)
Description: Only patient receiving treatment are considered as safety population.
Arm/Group | GRASPA (Non Allergic Population) | Reference L-asparaginase (Non Allergic Population) | GRASPA (Allergic Population)
All-Cause Mortality (participants affected / at risk) | 9/26 | 12/28 | 14/26
Serious Adverse Events (participants affected / at risk) | 23/26 | 26/28 | 23/26
Other Adverse Events (participants affected / at risk) | 26/26 | 28/28 | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GRASPA (Non Allergic Population) (N=26) | Reference L-asparaginase (Non Allergic Population) (N=28) | GRASPA (Allergic Population) (N=26)
Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (9) | 9 (9) | 7 (8)
drug hypersensitivity (Immune system disorders) | 3 (3) | 7 (7) | 3 (3)
Mucosal inflammation (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 5 (5)
lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 11 (23) | 7 (10) | 5 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 5 (9) | 4 (7)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 15 (15) | 8 (8) | 6 (6)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 4 (4) | 2 (2) | 0 (0)
Anal Abscess (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Septic shock (Infections and infestations) | 3 (3) | 1 (1) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Fusarium infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Human herpesvirus 6 infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GRASPA (Non Allergic Population) (N=26) | Reference L-asparaginase (Non Allergic Population) (N=28) | GRASPA (Allergic Population) (N=26)
Haematoma (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 7 (8) | 18 (21) | 17 (21)
Graft versus host disease (Immune system disorders) | 2 (2) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 2 (3) | 0 (0) | 4 (4)
Asthenia (General disorders) | 0 (0) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1)
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 2 (2)
Transaminases increased (Investigations) | 16 (40) | 16 (33) | 15 (21)
Hypokalaemia (Investigations) | 13 (13) | 11 (12) | 9 (12)
Antithrombin III decreased (Investigations) | 4 (7) | 20 (44) | 9 (11)
Gamma-glutamyltransferase increased (Investigations) | 8 (20) | 14 (15) | 7 (16)
Blood albumin decreased (Investigations) | 5 (5) | 11 (15) | 6 (7)
Hyponatraemia (Investigations) | 6 (6) | 10 (19) | 7 (8)
blood bilirubin increased (Investigations) | 4 (6) | 9 (11) | 7 (8)
Hyperglycaemia (Investigations) | 5 (6) | 7 (12) | 6 (12)
Activated partial thromboplastin time prolonged (Investigations) | 1 (2) | 4 (7) | 5 (5)
Hypocalcaemia (Investigations) | 3 (3) | 4 (4) | 1 (3)
Blood triglycerides increased (Investigations) | 2 (4) | 3 (4) | 3 (3)
Prothrombin level decreased (Investigations) | 0 (0) | 3 (5) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 2 (2) | 1 (1)
Blood potassium increased (Investigations) | 3 (3) | 2 (2) | 0 (0)
C-reactive protein increased (Investigations) | 2 (3) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 25 (76) | 27 (81) | 26 (74)
Thrombocytopenia (Blood and lymphatic system disorders) | 24 (69) | 26 (71) | 22 (71)
Neutropenia (Blood and lymphatic system disorders) | 24 (89) | 25 (93) | 25 (81)
Lymphopenia (Blood and lymphatic system disorders) | 21 (43) | 23 (43) | 20 (49)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 5 (17) | 7 (17) | 8 (13)
Hypofibrinogenaemia (Blood and lymphatic system disorders) | 9 (11) | 19 (37) | 11 (12)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (4) | 5 (9) | 3 (6)
Anaemia (Blood and lymphatic system disorders) | 7 (9) | 9 (14) | 6 (6)
Bone marrow failure (Blood and lymphatic system disorders) | 2 (2) | 3 (4) | 1 (1)
Blood phosphorus decreased (Blood and lymphatic system disorders) | 4 (5) | 3 (3) | 3 (3)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (3) | 2 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 1 (1) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 2 (2) | 6 (12) | 8 (9)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2)
renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Drug hypersensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 2 (3) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No